CLINICAL TRIAL: NCT00596544
Title: Sexual Functioning After Primary Treatment of Ovarian Cancer
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 04-124
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Ovarian Cancer; Sexual Dysfunction
Keywords: sexual dysfunction
MeSH Terms: conditions — Ovarian Neoplasms; Sexual Dysfunction, Physiological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: FSFI score <= 26
  Interventions: Behavioral: questionnaires
- 2: FSFI score >26
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — will be offered referral to the Sexual Health Clinic (SHC) at MSKCC for evaluation and possible treatment. The effectiveness and compliance of the intervention offered at the SHC will be assessed at approximately 3, 6 and 12 months using the FSFI, SAQ, CES-D, MSC and IES. At each evaluation they will complete a Health Surveillance Form (HSF). They will have completed the study at 12 months after entering the study or at the time they have evidence of recurrent disease requiring treatment
  Groups: 1
Behavioral: questionnaires — Those women who have a FSFI score > 26 will be reassessed at approximately 3, 6 and 12 months. They will complete the FSFI, SAQ, CES-D, IES, MSC and HSF at each assessment. They will be followed out until 12 months after entering the study or until they have evidence of recurrent disease.
  Groups: 2

SUMMARY:
The purpose of this study is to help us learn more about sexual problems after treatment for ovarian cancer. At this time, we do not know how many women have sexual problems after they are treated for ovarian cancer.

How common are sexual problems after treatment for ovarian cancer?

* What factors make women more likely to have sexual problems after treatment for ovarian cancer?
* What happens to sexual functioning over the first 12 months after treatment? ie.

Does it get better or worse?

• Does referral to a specialized sexual health clinic help?

ELIGIBILITY:
Inclusion Criteria:

* Women with any stage of invasive epithelial ovarian cancer who have completed frontline therapy within the past 6 months
* Women must have no clinical evidence of disease
* At least 18 years of age
* English speaking
* Able to participate in the informed consent process
* Women who present to Sexual Health Clinic for the first time and meet all other eligibility criteria are eligible. Their FSFI scores will be used to determine the primary endpoint of prevalence of sexual dysfunction. If they score over 26 on the FSFI, they may still elect to be followed at the SHC.

Exclusion Criteria:

* Active secondary cancer requiring cytotoxic chemotherapy at the time enrollment
* Evidence of recurrent/persistent disease by elevated CA125, findings on imaging (CT, PET scan etc) or physical examination
* Women with borderline (low malignant potential) ovarian cancers
* Women who are already in active evaluation and/or follow-up at the Sexual Health Clinic
* Women with a history of prior whole pelvic radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2004-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence of sexual dysfunction, as measured by Female Sexual Functioning Index (FSFI) among women who have completed first-line treatment for ovarian cancer within the last 6 months and currently have no evidence of disease. | conclusion of study

SECONDARY OUTCOMES:
To study the natural history of sexual functioning in women after primary treatment of ovarian cancer by using the FSFI at approximately 3, 6 and 12 months. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Jewell, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org